CLINICAL TRIAL: NCT03547843
Title: The Effects of Peer Co-led Educational Group Intervention for Adults With Attention-Deficit Hyperactivity/Impulsivity Disorder
Brief Title: The Effects of Peer Co-led Educational Group Intervention for Adults With Attention-Deficit Hyperactivity Disorder
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/2405 REK
Record Dates: First submitted 2018-04-25; First posted 2018-06-06 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Behavior therapy; Peer groups; Patient satisfaction; Feasibility studies
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Patient Satisfaction | interventions — Patient Education as Topic; Waiting Lists; Therapeutics

STUDY DESIGN:
Intervention Model Description: Pilot randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Experimental): Patients randomized to the intervention group will start with a group-based educational program immediately after the randomization.
  Interventions: Behavioral: Group-based education; Other: Standard treatment
- Waiting list (Active Comparator): Participants randomized to the waiting list control group receive no educational intervention for the duration of the 10 weeks. During this period participants can receive standard treatment, consisting of diagnostic treatment with medication.
  Interventions: Behavioral: Waiting list; Other: Standard treatment

INTERVENTIONS:
Behavioral: Group-based education — The group-based educational program consists of two sessions that run over two consecutive weeks. Each session consists of a lecture from a recruited expert on the topic of the session and by expert patients with a following discussion of the topic facilitated by the course leader.
  Other Names: Patient education
  Arms: Educational intervention
Behavioral: Waiting list — No educational intervention for the duration of the 10 weeks. During this period participants can receive standard treatment.
  Arms: Waiting list
Other: Standard treatment — Diagnostic treatment with medication. In addition, some patients receive cognitive behavioral therapy (not systematically given to every patient). If needed, patients are also offered assistance with regard to economy, housing, education, and work as well as contact with family and network.
  Other Names: Treatment as usual

SUMMARY:
Peer co-led education describes educators who are expert patients, user representatives or former patients, participating and teaching in educational interventions in cooperation with health care professionals. Peer co-led education is included in the Norwegian national guidelines for treatment of mental disorders, but despite some promising results for the treatment of other conditions, still little is known about the efficacy of peer co-led educational group interventions interventions for adults with attention deficit and hyperactivity disorder (ADHD).

This pilot trial will evaluate patient satisfaction with and preliminary efficacy of a 2-session peer co-led educational group program designed to address specific challenges faced by adults diagnosed with ADHD at an outpatient clinics in mid-Norway.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ADHD-diagnosis
* speaking a Scandinavian language

Exclusion Criteria:

* Unable to give informed consent
* Psychosis
* Severe learning difficulties

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in client Satisfaction | from baseline to 2-weeks follow-up
  Client satisfaction will be measured with Client Satisfaction Questionnaire, short form (Attkisson & Zwick, 1982). The scale consists of 8 items scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction). Total scores range from 8 to 32, with higher scores indicating greater satisfaction.
change in patient activation | from baseline to 10-weeks follow-up
  Patient activation will be measured with the Norwegian version of the Patient Activation Measure Mental Health (PAM-MH) (Green et al 2010))

SECONDARY OUTCOMES:
change in general self-efficacy | from baseline to 10 weeks follow-up
  General Self-Efficacy Scale, 6-item scale ranging from 1 ('not at all true') to 4 ('exactly true'). Total scores range from 6 to 24, with higher scores indicating greater self-efficacy. (Romppel et al 2013)
change in ADHD-related symptoms | from baseline to 10 weeks follow-up
  Hopkin's Symptom Checklist (SCL), 9-items scale with high scores on SCL-9 indicating ADHD-related symptom burden (Eich et al 2011)
change in ADHD-related symptoms | from baseline to 10 weeks follow-up
  Norwegian version of the WHO Adult ADHD Self-report scale, ASRS Short Form (Kessler et al 2005)
change in Quality of Life | from baseline to 10 weeks follow-up
  Adult Attention Deficit/Hyperactivity Disorder Quality of Life Scale, AAQoL short Form (Brod et al 2006)

OTHER OUTCOMES:
Use of health services and work participation | through study completion, an average of 24 weeks
  Self-reported work participation and received services: 3 questions about both work status and received treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Løvaas, md phd, Study Director — St. Olavs Hospital
Locations (1):
- Tiller DPS, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skliarova T, Grawe RW, Vaag J, Mandahl A, Kolltveit I, Lovas I, Torgersen T, Lara-Cabrera ML. Pilot randomised controlled trial on the feasibility and intervention satisfaction with an educational group programme for adults with attention deficit hyperactivity disorder and their caregivers. BMC Psychiatry. 2025 Feb 20;25(1):161. doi: 10.1186/s12888-025-06570-4. PMID 39979888